CLINICAL TRIAL: NCT03381599
Title: Quantification and Qualification of Stem Cells After Peripheral Mobilization and Harvest for Orthopaedic Point of Care Application
Brief Title: Stem Cells After Peripheral Mobilization and Harvest
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: Auburn University (Other); Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16398
Record Dates: First submitted 2017-12-14; First posted 2017-12-22 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Stem Cells; Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone marrow aspirate (Experimental): This study will utilize one group of participants. This group of participants will have bone marrow aspirate and a blood sample collected from the iliac crest and subsequently analyzed with the Arthrex Angel system. Thirty days following bone marrow aspiration, participants will receive a subcutaneous Filgrastim injection on four serial days. On the fifth day, a peripheral blood sample sample will be obtained.
  Interventions: Drug: Filgrastim Injection

INTERVENTIONS:
Drug: Filgrastim Injection — Filgrastim of 10 ug/kg/day will be given for four serial days.
  Other Names: Neupogen

SUMMARY:
The proposed study is a controlled laboratory study where stem cell content of bone marrow aspirate will be compared prior to and following pharmaceutical mobilization. Participants who meet the inclusion/exclusion criteria will have a bone marrow sample taken from the iliac crest. The sample will be tested to determine stem cell content and for the presence of proteins which are of interest in orthopedic treatments. Thirty days following the baseline bone marrow collection, participants will receive a subcutaneous injection of Filgrastim daily for four serial days. On the fifth day, a peripheral blood sample will be taken and processed.

DETAILED DESCRIPTION:
Orthopaedic practitioners have begun to augment surgical procedures and treat degenerative conditions, such as osteoarthritis, with injections of bone marrow aspirate. Clinical application studies have suggested that success is dependent upon the number of stem cells harvested and utilized. Pharmaceutical mobilization, with agents such as Filgrastim (Neupogen), followed by peripheral harvest of stem cells has supplanted bone marrow aspirate for hematologic oncologic clinical practice of stem cell transplant, with established safety and efficacy.

The proposed study is a controlled laboratory study where stem cell content of bone marrow aspirate will be compared prior to and following pharmaceutical mobilization using Filmgrastim (Neupogen). Participants will undergo a screening examination consisting of a physical examination and blood work. A standard venipuncture will be performed in the left or right arm and a 5.0 mL vacationer tube will be filled with blood and a 60 mL syringe pre-filled with anticoagulant will be filled with blood. The blood will be analyzed with flow cytometry, a histologic smear, a complete blood count (CBC) with white blood cell (WBC) differential, and chemokine/cytokine analyst with ELISA testing. The blood in the 60.0 mL syringe will be processed with the Arthrex Angel system. The buffy coat component of the blood will be analyzed.

On a separate day, participants who meet the inclusion/exclusion criteria will have a bone marrow sample taken from the iliac crest. The participant will lay on their side and 20 mL of 1% lidocaine will be injected into the anticipated incision site. A 1 cm incision in the skin, advancing a trotter into the bone marrow cavity, aspirating 5 cc of bone marrow with a 5 mL syringe and placement of the sample into a 5 mL vaccutainer syringe, and filling a 60.0 ml syringe pre-filled with 8 ml of citrate anticoagulant with bone marrow aspirate. The bone marrow in the 5 mL vaccutainer will be analyzed by flow cytometry, a histologic smear, a CBC with WBC differential, and chemokine/cytokine analysis with ELISA testing. The bone marrow in the 60.0 mL syringe will be processed with the Arthrex Angel system. The sample will be tested to determine stem cell content and for the presence of proteins which are of interest in orthopedic treatments.

Thirty days following the baseline bone marrow collection, participants will receive a subcutaneous injection of Filgrastim daily for four serial days. A blood sample of 5 mL will be collected each day of the injection to obtain a CBC and WBC differential. On the fifth day, a peripheral blood sample will be taken and processed following the same procedures as the first sample.

It is hypothesized that with a pharmaceutical mobilization method and the Arthrex Angel system, clinicians can harvest more stem cells than with bone marrow aspiration alone.

ELIGIBILITY:
Inclusion Criteria:

* Weight 110-220 pounds
* Healthy

Exclusion Criteria:

* Previous allergic reaction to Filgrastim, lidocaine, or other injectable numbing agent
* White blood count greater than 20,000/mcL
* Latex allergy
* Diabetes
* Any autoimmune disorder
* Any blood disorder requiring immunosuppression
* Cancer
* Ongoing infectious disease
* Significant cardiovascular, renal, hepatic, or pulmonary disease
* Sickle cell or other blood disorders
* Presence of abdominal tenderness with palpation upon physical examination
* Signs of splenomegaly upon physical examination
* Abnormal lung fields upon physical examination

Ages: 19 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Change in Stem Cell Count | Baseline to Day 32
  Quantity and quality of the harvested stem cells

SECONDARY OUTCOMES:
Complete blood count | Day 1, Day 2, Day 28, Day 29, Day 30, Day 31 Day 32
  Participants white blood cell count/differential
Chemokine/Cytokine | Day 1, Day 2, Day 28, Day 29, Day 30, Day 31 Day 32
  Participants chemokine/cytokine count

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Anz, MD, Principal Investigator — Andrews Research & Education Foundation; Michael Goodlett, MD, Study Director — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03381599/Prot_SAP_ICF_000.pdf